CLINICAL TRIAL: NCT00576563
Title: Rectal Cancer: Determination of the Predictive Value by Use of FDG-PET-CT Scans and Blood Proteins for the Prognosis of Patients With Rectal Cancer
Brief Title: Rectal Study: Value of Repeated FDG-PET-CT Scans in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-02
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Rectum Cancer
Keywords: rectal cancer; blood proteins; irradiation; FDG-PET-CT
MeSH Terms: conditions — Rectal Neoplasms | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG PET CT (Other): To investigate the evolution of the 18F-deoxyglucose (FDG) uptake and the tumour characteristics determined in the plasma of patients with rectal cancer during and after radiotherapy or combined radiotherapy and chemotherapy.
  Interventions: Drug: FDG

INTERVENTIONS:
Drug: FDG — contrast medium
  Other Names: Omnipaque 350/ 18 Fluor FDG

SUMMARY:
To investigate the evolution of the 18F-deoxyglucose (FDG) uptake and the tumour characteristics determined in the plasma of patients with rectal cancer during and after radiotherapy or combined radiotherapy and chemotherapy.

The changes of the FDG uptake of the primary tumour and the evolution of key tumour characteristics during radiotherapy alone or in combination with chemotherapy will be predictive for the pathological tumour response.

Study hypothesis The changes of the FDG uptake of the primary tumour and the evolution of key tumour characteristics during radiotherapy alone or in combination with chemotherapy will be predictive for the pathological tumour response.

DETAILED DESCRIPTION:
This translational research part is aiming to give more insights in the way radiation injury and tumour response develops.

It involves three parts:

1. Repetitive FDG-PET-CT scans in order to assess early tumour response monitoring.
2. Blood sampling before, during and after radiotherapy in order to find predictors for normal tissue injury and for tumour response.
3. Extra staining of tumour biopsies.

1. FDG-PET-CT scans The FDG-PET-CT scan with i.v. contrast gives information of the tumour metabolism and its morphology. The pre-treatment max SUV is prognostic as a high value confers a worse prognosis. Our group showed both in vitro and in vivo that a high FDG uptake is due to tumour hypoxia. The evolution of the max SUV during radiotherapy may thus be predictive for the ultimate tumour response. Therefore, two extra FDG-PET-CT scans will be done during radiotherapy for the group of patients receiving long-term radiochemotherapy: one at day 7 and one at day 14. This will enable calculation of the max SUV kinetics during treatment. Tumour response will be determined by FDG-PET-CT scans 3-5 days after the short- course of radiotherapy or 6-8 weeks after the long- term radiochemotherapy.

2 Blood samples Blood collection and processing before, during and after radiotherapy will be done according to the serum protocol. For performing ELISA's blood samples should be collected and put in the freezer. The analysis of all blood material will be performed months to years after collection and re-analysis with regard to the described protein groups may be necessary depending on the outcome.

1. Before radiotherapy, 10 millilitres of blood will be taken.
2. At day 7, day 14 and 6-8 weeks after the end of radiotherapy for the long- term radiotherapy or 3-5 days after the short - course of radiotherapy,i.e. at the same days that the FDG-PET-CT scans will be performed, 10 millilitres serum (EDTA tube) will be taken to investigate the evolution of the proteins during and after treatment, for its kinetics may be important as predictive factors.

3 Extra staining of tumour biopsies The tumour biopsies may be stained with markers for proliferation (e.g. KI 67), apoptosis (e.g. M30), hypoxia (e.g. HIF, CA 9, Glut 1 and 3) and others (e.g. EGFR and EGFRvIII), in order to correlate these measurements with response.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven rectal cancer
* UICC stage I-IV
* WHO performance status 0-2
* Less than 10 % weight loss in the last 6 months
* In case of previous chemotherapy, radiotherapy can start after a minimum of 21 days after the last chemotherapy course
* No recent (< 3 months) severe cardiac disease (arrhythmia, congestive heart failure,infarction)
* Life expectancy more than 6 months
* Measurable cancer
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant and willing to take adequate contraceptive measures during the study
* Have given written informed consent before patient registration
* No previous radiotherapy to the pelvis

Exclusion Criteria:

* Not adenocarcinoma histology
* History of prior pelvis radiotherapy
* Recent (< 3 months) myocardial infarction
* Uncontrolled infectious disease
* Less than 18 years old
* Pregnant or not willing to take adequate contraceptive measures during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-03; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The metabolic tumour response by PET scan will be determined according to the EORTC criteria (appendix 1)61. The pathological tumour response will be determined according to Dworak and Wheeler.62,63 | 5 years

SECONDARY OUTCOMES:
Clinical examination(weight, performance status including the CTCv3.0 scale for acute and late reactions) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Lammering, MD PHD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands